CLINICAL TRIAL: NCT02509611
Title: Effects of Yoga on Redox Status, Motor Function and Psychosocial Well-being in Individuals With Parkinson's Disease
Brief Title: Effects of Yoga on Parkinson's Disease
Acronym: HYPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1506M74261
Record Dates: First submitted 2015-07-20; First posted 2015-07-28 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2017-06

CONDITIONS: Parkinson's Disease
Keywords: Yoga; Parkinson's disease; redox status; motor function
MeSH Terms: conditions — Parkinson Disease | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate treatment (Experimental): Participants who are randomly assigned to the immediate treatment group will receive 60-minute biweekly Hatha yoga for 12 weeks.
  Interventions: Other: Hatha yoga
- Waitlist control (Active Comparator): Participants who are randomly assigned to the wait-list group will receive no intervention during the first 12 weeks. Not only will they serve as the comparative group, they will also serve as their own control and receive the same yoga intervention at the end of 12 weeks when the immediate treatment group completed their program.
  Interventions: Other: Hatha yoga

INTERVENTIONS:
Other: Hatha yoga — Yoga programs that were used in previous PD studies will be incorporated into the design of the proposed intervention program. Two yoga experts who are specialized in musculoskeletal/neurological disorders will review the program. The yoga intervention classes will be taught by a Registered Yoga Teacher. The 60 minute long yoga session will be held twice a week for 12 weeks at a community center in St. Louis Park.
  Other Names: Yoga

SUMMARY:
The study's purpose is to assess the effect of yoga on measures of oxidative stress (i.e. reduction-oxidation [redox] status); motor function; and psychosocial well-being, and the feasibility and acceptability of implementing a Hatha yoga program in PD subjects.

DETAILED DESCRIPTION:
The specific aims of this study are:

Aim 1: Determine the effect of a 12-week Hatha yoga program on redox status in individuals with PD.

Hypothesis 1a: Participants in the intervention group will have greater increases in total GSH levels and GSH: GSSG ratios from baseline than participants in the wait-list control group.

Hypothesis 1b: Compared to pre-intervention, wait-list participants will have higher total GSH levels and GSH: GSSG ratios after receiving the intervention.

Aim 2: Examine the effect of a 12-week Hatha yoga program on motor function (gait, balance, strength, flexibility, and physical activity level) and psychosocial well-being (mood, cognitive function, sleep quality, QoL) in individuals with PD.

Hypothesis 2a: Participants in the intervention group will have greater improved scores on the motor Unified Parkinson's Disease Rating Scale (UPDRS), range of motion (ROM), biomechanical force platforms tests, Beck Depression Inventory (BDI), Parkinson's Disease Sleep Scale (PDSS), Parkinson's Disease Quality of Life Questionnaire (PDQUALIF), and Montreal Cognitive Assessment than wait-list participants.

Hypothesis 2b: Compared to pre-intervention, wait-list participants will have improved scores on the motor UPDRS, ROM, biomechanical force platforms tests, BDI, PDSS, and PDQUALIF after receiving the intervention.

Aim 3: Determine the feasibility and acceptability of Hatha yoga program for PD subjects, and fidelity of the yoga program.

Hypothesis 3: The program retention rate will be > 70%, the average attendance rate will be > 70% per class, and no yoga related adverse events will be reported during the study. Most participants will react positively to the yoga program.

Methods Design and Sample A randomized controlled trial design with two groups will be used: a treatment group (n=10) and a wait-list control group (n=10). After randomization, participants in the treatment group will receive 60-minute biweekly Hatha yoga for 12 weeks, and participants in the wait-list group will receive no intervention. Wait-list participants will also serve as their own control and receive the same yoga intervention at the end of 12 weeks when the treatment group completed their program. Participants will be recruited from clinics via flyers, and through local and national PD networks.

Yoga programs that were used in previous PD studies will be incorporated into the design of the proposed intervention program. 19, 31, 32 Two yoga experts who are specialized in musculoskeletal/neurological disorders will review the program. The yoga intervention classes will be taught by a Registered Yoga Teacher. Classes will be held at a community center in St. Louis Park.

Resting blood samples will be collected at the Clinical Translational Science Institute (CTSI) facility by a trained phlebotomist and total GSH and redox status analyzed by a co-investigator. Biomechanical assessment and survey data will be collected in the Konczak laboratory by a trained graduate research assistant. All data will be collected at baseline and 12 weeks from both treatment and wait-list control groups. The 12 weeks data from the wait-list participants will serve as their second baseline before they began the intervention program. Their post intervention data will be collected at 24 weeks post randomization to increase power.

Study Endpoints:

1. Primary endpoint: redox status at 12 weeks.
2. Secondary endpoint: motor function (gait, balance, strength, flexibility, physical activity level) and psychosocial well-being (mood, cognitive function, sleep quality, QoL) at 12 weeks.
3. Tertiary endpoint: yoga feasibility, acceptability, and program fidelity. The sample size of 20, with attrition rate of 20%, has 78% power to detect an effect size of 1.0 when comparing the change before and after the yoga intervention. Both between groups and within group comparisons will be conducted. Descriptive statistics will be used to analyze and report demographic, feasibility, and acceptability data. Inferential statistics (t-test or non-parametric equivalent such as Mann-Whitney, and chi-square test) will be used to analyze the objective and subjective outcomes of Aims 1 & 2. The α level will be set at ≤ .05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with idiopathic PD;
* On optimized dopaminergic therapy for 4 weeks prior to enrollment; and
* Have not practiced any form of yoga regularly (more than 2 days a week) in the past 6 months; and
* Not currently participating in a supervised exercise program more than 2 days a week

Exclusion Criteria:

* Atypical Parkinsonism or other significant brain conditions such as a stroke;
* Fell more than once in the past 3 months;
* Moderate to severe cognitive impairment (scored <26) as indicated by the Montreal Cognitive Assessment;
* Decline in immune function such as pneumonia or systemic infection;
* Spinal fusion or other orthopedic surgery in the past 6 months;
* Unstable cardiovascular conditions;
* Significant mental disease or psychosis;
* Not able to ambulate 6 meters steadily without assistive device.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Redox status | 12 weeks
  The antioxidant glutathione (GSH) and the GSH: glutathione disulfide (GSSG) ratio will be measured at baseline and at the end of the program.

SECONDARY OUTCOMES:
Motor function | 12 weeks
  Gait and strength will be measured using motor Unified Parkinson's Disease Rating Scale (UPDRS) biomechanical force platforms tests: Force plate system (OR6-5 AMTI) - 2D sway path length of center of mass during 20s standing.
Motor function | 12 weeks
  Balance will be measured using the motor UPDRS and biomechanical force platforms tests: Force plate system (OR6-5 AMTI) - range of anterior-posterior and medial-lateral away, total sway area, and duration of one-legged stance.
Motor function | 12 weeks
  Flexibility will be evaluated by measuring range of motion using a goniometer.
Cognitive function | 12 weeks
  Cognitive function will be evaluated using the Montreal Cognitive Assessment test.
Mood | 12 weeks
  Mood will be evaluated using the Beck Depression Inventory scale.
Sleep quality | 12 weeks
  Sleep quality will be evaluated using the Parkinson's Disease Sleep Scale.
Physical activity level | 12 weeks
  Longitudinal Aging Study Amsterdam scale will be used to evaluate physical activity levels in PD subjects.
Quality of Life | 12 weeks
  Parkinson's Disease Quality of Life Questionnaire will be used.

OTHER OUTCOMES:
Yoga feasibility | Baseline and 12 weeks
  Number of eligible subjects, total average number of class attendance, number and type of yoga related adverse events, and retention rate.
Yoga acceptability | 12 weeks
  A short questionnaire will be used to evaluate participants' self-report satisfaction with the yoga program, perceived appropriateness of the program, and intention to continue use of the program.
Yoga program fidelity | 4 weeks, 8 weeks, and 12 weeks
  The PI will evaluate the accuracy/consistency of the intervention program.

CONTACTS AND LOCATIONS:
Overall Officials: Corjena Cheung, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886